CLINICAL TRIAL: NCT02115529
Title: A Randomized Controlled Trial of Cesamet(R) (Nabilone) for the Prevention of Postoperative Nausea and Vomiting in Elective Surgery
Brief Title: Study of Prevention of Postoperative Nausea and Vomiting Using Cesamet
Acronym: Cesamet
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 13-242
Record Dates: First submitted 2014-03-03; First posted 2014-04-16 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-11

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — nabilone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cesamet (nabilone) (Active Comparator): 0.5 mg capsule containing Cesamet (single dose) given preoperatively
  Interventions: Drug: Nabilone
- Placebo (Placebo Comparator): identical capsule containing placebo (single dose) given preoperatively
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nabilone — Nabilone (0.5 mg) or placebo given preoperatively
  Other Names: Cesamet
  Arms: Cesamet (nabilone)
Drug: Placebo — Placebo Comparator: identical capsule containing placebo (single dose) given preoperatively
  Arms: Placebo

SUMMARY:
Untreated, one third of patients undergoing general anesthesia will have postoperative nausea, vomiting, or both.

Patients often rate postoperative nausea and vomiting (PONV) as worse than postoperative pain. PONV increases the risk of aspiration and has been associated with suture dehiscence, esophageal rupture, subcutaneous emphysema, and bilateral pneumothoraxes. PONV frequently delays discharge, and is the leading cause of unexpected hospital admission after planned ambulatory surgery.

Nabilone (Cesamet®) is a synthetic cannabinoid developed in the 1970s which is a potent CB1 agonist. The use of nabilone in preventing nausea and vomiting in patients receiving chemotherapy has been thoroughly investigated. Results from clinical studies demonstrated the efficacy, safety, and tolerability of Cesamet in this population. There has been success in the past translating treatments for chemotherapy-induced nausea and vomiting (ie. 5-HT receptor agonists including Ondansetron and Granisetron) to use in the perioperative environment.

Only one RCT has studied the use of nabilone for the reduction of PONV. Published in 1995, this study compared the administration of either Cesamet 2 mg or metoclopramide 10 mg given 90 minutes before the operation in patients scheduled for elective hysterectomy in 60 women. This study failed to show any significant difference between groups. There are several limitations to this study including a poorly optimized dosing regimen, a small sample size, and a comparison group lacking clinical generalizability.

This study will investigate the use Cesamet vs Placebo, in addition to the regular antiemetic treatment which patients receive at the discretion of the managing anesthesiologist, for the prevention of PONV. The study group will include patients undergoing general anesthesia for elective ambulatory surgery with at least 3 risk factors (>60% risk) for the development of PONV.

DETAILED DESCRIPTION:
See above

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older with an American Society of Anesthesiologists (ASA) physical status of I to III who are scheduled to undergo elective surgery under general anesthesia with pre-anesthesia consultation prior to surgery.
* Subjects must be able to swallow study medication;
* At a risk of postoperative nausea and vomiting of at least 61% percent, according to a simplified risk score, based on the presence of at least three of the following risk factors: female sex, nonsmoker status, anticipated use of postoperative opioid and previous PONV or motion sickness.

Exclusion Criteria:

* Subjects with clinically significant or unstable cardiac, respiratory, hepatic, renal, or other major organ system disease
* Patients who will not be admitted to the PACU post-operatively (patients who are immediately transferred to the ICU)
* Known sensitivity to marijuana or other cannabinoid agents
* Psychotic illness or depression
* Addiction to illicit substances or alcohol
* Non-psychotic emotional disorders.
* Pregnant or lactating
* Subjects who suffer from chronic nausea and/or vomiting;
* Has had treatment with any other investigational drug within 12 weeks prior to randomization
* Subjects who, in the opinion of the investigator, would experience an unacceptable risk from administration of study drug

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 331 (Actual)
Dates: Start 2014-04; Primary Completion 2015-01 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative nausea and/or vomiting | Prior to discharge from postanesthesia care unit, an expected average of two hours

SECONDARY OUTCOMES:
Number of antiemetic rescue medications given postoperatively. | Prior to discharge from postanesthesia care unit, an expected average of two hours

OTHER OUTCOMES:
Standardized score of nausea and/or vomiting severity if PONV occurs. | Prior to discharge from postanesthesia care unit, an expected average of two hours
Pain score during the immediate post-operative period. | Prior to discharge from postanesthesia care unit, an expected average of two hours
Use of intraoperative and postoperative opioids | Prior to discharge from postanesthesia care unit, an expected average of two hours
Rates of known side effects. | Prior to discharge from postanesthesia care unit, an expected average of two hours
  Nabilone side effects include: drowsiness, vertigo, psychological high, dry mouth, depression, blurred vision, sensation disturbance, anorexia, headache, euphoria, and hallucinations (based on patient self-reporting).
Time to discharge from the PACU. | Prior to discharge from postanesthesia care unit, an expected average of two hours
Rates of admission due to PONV | Prior to discharge from postanesthesia care unit, an expected average of two hours
Antiemetics given prophylactically by the anesthesiologist. | Until discharge from postanesthesia care unit, an expected average of two hours

CONTACTS AND LOCATIONS:
Overall Officials: Aaron P Hong, MD, FRCPC, Principal Investigator — St Michael's Hospital, University of Toronto
Locations (1):
- St Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Habib AS, Gan TJ. Evidence-based management of postoperative nausea and vomiting: a review. Can J Anaesth. 2004 Apr;51(4):326-41. doi: 10.1007/BF03018236. PMID 15064261
- [Background] Weinstein RS. Glucocorticoid-induced osteonecrosis. Endocrine. 2012 Apr;41(2):183-90. doi: 10.1007/s12020-011-9580-0. Epub 2011 Dec 15. PMID 22169965
- [Background] Pertwee RG. Receptors and channels targeted by synthetic cannabinoid receptor agonists and antagonists. Curr Med Chem. 2010;17(14):1360-81. doi: 10.2174/092986710790980050. PMID 20166927
- [Background] Ware MA, Daeninck P, Maida V. A review of nabilone in the treatment of chemotherapy-induced nausea and vomiting. Ther Clin Risk Manag. 2008 Feb;4(1):99-107. doi: 10.2147/tcrm.s1132. PMID 18728826
- [Background] Hsu ES. A review of granisetron, 5-hydroxytryptamine3 receptor antagonists, and other antiemetics. Am J Ther. 2010 Sep-Oct;17(5):476-86. doi: 10.1097/MJT.0b013e3181ea7821. PMID 20844345
- [Background] Lewis IH, Campbell DN, Barrowcliffe MP. Effect of nabilone on nausea and vomiting after total abdominal hysterectomy. Br J Anaesth. 1994 Aug;73(2):244-6. doi: 10.1093/bja/73.2.244. PMID 7917745
- [Background] Koivuranta M, Laara E, Snare L, Alahuhta S. A survey of postoperative nausea and vomiting. Anaesthesia. 1997 May;52(5):443-9. doi: 10.1111/j.1365-2044.1997.117-az0113.x. PMID 9165963
- [Background] Gan TJ. Postoperative nausea and vomiting--can it be eliminated? JAMA. 2002 Mar 13;287(10):1233-6. doi: 10.1001/jama.287.10.1233. No abstract available. PMID 11886298
- [Background] Apfel CC, Korttila K, Abdalla M, Kerger H, Turan A, Vedder I, Zernak C, Danner K, Jokela R, Pocock SJ, Trenkler S, Kredel M, Biedler A, Sessler DI, Roewer N; IMPACT Investigators. A factorial trial of six interventions for the prevention of postoperative nausea and vomiting. N Engl J Med. 2004 Jun 10;350(24):2441-51. doi: 10.1056/NEJMoa032196. PMID 15190136
- [Background] Bremner WG, Kumar CM. Delayed surgical emphysema, pneumomediastinum and bilateral pneumothoraces after postoperative vomiting. Br J Anaesth. 1993 Aug;71(2):296-7. doi: 10.1093/bja/71.2.296. PMID 8123411
- [Background] Fortier J, Chung F, Su J. Unanticipated admission after ambulatory surgery--a prospective study. Can J Anaesth. 1998 Jul;45(7):612-9. doi: 10.1007/BF03012088. PMID 9717590
- [Background] Macario A, Weinger M, Carney S, Kim A. Which clinical anesthesia outcomes are important to avoid? The perspective of patients. Anesth Analg. 1999 Sep;89(3):652-8. doi: 10.1097/00000539-199909000-00022. PMID 10475299
- [Background] Product monograph, Nabilone (Nabilone), submission control no: 124406, Valeant Canada Limitée/Limited, March 17, 2009
- [Derived] Levin DN, Dulberg Z, Chan AW, Hare GM, Mazer CD, Hong A. A randomized-controlled trial of nabilone for the prevention of acute postoperative nausea and vomiting in elective surgery. Can J Anaesth. 2017 Apr;64(4):385-395. doi: 10.1007/s12630-017-0814-3. Epub 2017 Feb 3. PMID 28160217